CLINICAL TRIAL: NCT03088917
Title: 'Fibrosis in the Lost Hepatitis C Population - Track, Trace and Treat' A Prospective Cohort Study Assessing the Impact of Loss to Follow-up on Liver Fibrosis in Chronic Hepatitis C.
Brief Title: 'Fibrosis in the Lost Hepatitis C Population - Track, Trace and Treat'
Acronym: Track&Trace
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joost Drenth, Professor, MD, PhD, Radboud University Medical Center
Other Study IDs: 2017-3198
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum samples will be saved in the biobank after participation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lost to follow-up patients: This so-called lost population consists of all patients, that in the past have been diagnosed with hepatitis C at the Radboudumc but who are currently lost to or have been withdrawn from follow-up. The time-span of interest will be 2000-2015.

SUMMARY:
Objective:

To coordinate active tracing of chronic hepatitis C patients lost to follow-up to inform them about there disease severity and treatment options.

Study design: This is a prospective cohort study, which will start as a pilot study in the Radboudumc Population: lost to follow-up chronic hepatitis C patients in the region Nijmegen. This so-called lost population consists of all patients, that in the past have been identified at the Radboudumc but who are currently lost to or have been withdrawn from follow-up. The time-span of interest will be 2000-2015. We estimate that this project will retrace 100 lost patients through this search.

ELIGIBILITY:
Inclusion Criteria:

* ever diagnosed with hepatitis C, lost to follow-up

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lost to follow-up chronic hepatitis C patients in the region Nijmegen. This so-called lost population consists of all patients, that in the past have been diagnosed with hepatitis C at the Radboudumc but who are currently lost to or have been withdrawn from follow-up. The time-span of interest will be 2000-2015.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joost Drenth, Md,PhD,Prof, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Possibly individual data on primary and secondary outcomes can be requested from reserachers or shared via digital research environment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After identification of lost to follow-up hepatitis C patients, patients who were alive and residing in the Netherlands were invited for re-evaluation at the outpatient clinic.
Pre-assignment Details: After invitation, patients could not be enrolled (defined as the signing of informed consent) for multiple reasons. These reasons are described below.
Groups:
- Invited Lost to Follow-up Patients: Alive patients who were anti-HCV and/or HCV RNA positive in the period 2000-2015 who have not been treated and were residing in the Netherlands, were invited for re-evaluation at the outpatient clinic.
Period: Overall Study
Arm/Group | Invited Lost to Follow-up Patients
Started | 106
Completed | 10
Not Completed | 96
Not completed — In care/cured elsewhere | 15
Not completed — Refuse re-evaluation | 13
Not completed — Contact not established | 13
Not completed — Severe comorbidity/short life expectancy | 5
Not completed — Moved outside study region | 50

BASELINE CHARACTERISTICS:
Groups:
- Re-evaluated Lost to Follow-up Patients: Invited lost to follow-up patients who were seen at the outpatient clinic.
Arm/Group | Re-evaluated Lost to Follow-up Patients
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [58 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 10
Country of birth [Count of Participants; unit: Participants]
  Netherlands | 8
  England | 1
  France | 1
HCV transmission route [Count of Participants; unit: Participants]
  Intravenous drug use | 7
  Blood transfusion | 3
Years since last hospital contact [Median (Full Range); unit: years] | 13.5 [1 to 20]
Treatment experienced [Count of Participants; unit: Participants] — Defined as having any (previously) registered HCV treatment, e.g. (pegylated) interferon or direct acting antivirals, with or without ribavirin
  Participants | 5
RNA-positive [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Liver Fibrosis Stage
Description: Fibrosis stage according to elastography (liver stiffness in kPa) and/or liverbiopsy (staging according to Metavir). Stage F0/1 equals minimal fibrosis, stage F2 equals significant fibrosis and stage F3/F4 equals advanced fibrosis (including cirrhosis). For elastography, F0/1 is defined as liver stiffness <7.1 kPa, F2 as liver stiffness between 7.1 and 9.4 kPa and F3/F4 as liver stiffness >9.4 kPa. For liver biopsy, F0/1 is defined as the presence of no fibrosis or minimal fibrosis without the presence of septa, F2 as the presence of portal fibrosis with a few septa and F3/F4 as the presence of septal fibrosis or cirrhosis. The higher the fibrosis stage, the worse the outcome.
Time Frame: Baseline
Population: Liver fibrosis was only assessed in patients who were HCV RNA-positive at baseline, i.e. in 5 out of a total of 10 re-evaluated patients.
Measure: Count of Participants; unit: Participants
Groups:
- RNA-positive Re-evaluated Lost to Follow-up Patients: LTFU patients who were still RNA-positive at the re-evaluation visit.
Arm/Group | RNA-positive Re-evaluated Lost to Follow-up Patients
Number analyzed (Participants) | 5
Participants
  F0/1 (<7.1 kPa) | 3
  F2 (7.1 - 9.4 kPa) | 1
  F3/F4 (>9.4 kPa) | 1

2. Secondary Outcome: Reasons for Loss to Follow-up
Description: through chart review or questioning screening event
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Re-evaluated Lost to Follow-up Patients
Number analyzed (Participants) | 10
Participants
  Patient: therapy refusal/contra-indication/no-show | 2
  Therapy-related: no indication or options | 2
  Care-related: no adequate follow-up planned | 5
  Unknown | 1

3. Secondary Outcome: Genotype Distribution
Description: Genotype distribution among RNA-positive patients
Time Frame: Baseline
Population: HCV genotype was only determined in patients who were HCV RNA-positive at baseline, i.e. 5 out of a total of 10 re-evaluated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | RNA-positive Re-evaluated Lost to Follow-up Patients
Number analyzed (Participants) | 5
Participants
  1a | 2
  1b | 2
  3a | 1

4. Secondary Outcome: Fibrosis Progression
Description: Fibrosis stage comparison in patients with a previously recorded fibrosis measurement, either with Fibroscan or liver biopsy. This previous measurement will be compared to the result of the Fibroscan performed during re-evaluation.
Time Frame: Baseline
Population: Fibrosis progression could only be measured if patients had a previous fibrosis measurement, either by liver biopsy or liver stiffness measurement. This was the case in 3 out of 5 HCV RNA-positive patients, or 3 out of 10 re-evaluated patients.
Measure: Count of Participants; unit: Participants
Groups:
- RNA-positive Re-evaluated Lost to Follow-up Patients: RNA-positive patients with a previous fibrosis measurement.
Arm/Group | RNA-positive Re-evaluated Lost to Follow-up Patients
Number analyzed (Participants) | 3
Participants
  No progression (F0/1 stayed F0/1) | 2
  Progression (F0/1 became F4) | 1

5. Secondary Outcome: Treatment Outcome
Description: Sustained virological response in treated patients, defined as non-detectable HCV RNA at least 12 weeks after end of treatment
Time Frame: At least 12 weeks after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RNA-positive Re-evaluated Lost to Follow-up Patients
Number analyzed (Participants) | 5
Participants
  Elbasvir/grazoprevir 12 weeks | 2
  Glecaprevir/pibrentasvir 8 weeks | 2
  Sofosbuvir/velpatasvir 12 weeks | 1

ADVERSE EVENTS:
Time Frame: Full duration of treatment: 8 or 12 weeks.
Description: Adverse events could only be reported in treated patients. Only 5 out of 10 re-evaluated patients were HCV RNA-positive and therefore only 5 had to be treated. Adverse events for these 5 patients are presented.
Groups:
- Treated Patients: RNA-positive patients who received treatment with interferon-free direct antiviral regimens.
Arm/Group | Treated Patients
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03088917/Prot_SAP_000.pdf